CLINICAL TRIAL: NCT02799602
Title: A Randomized, Double-blind, Placebo Controlled Phase III Study of Darolutamide (ODM-201) Versus Placebo in Addition to Standard Androgen Deprivation Therapy and Docetaxel in Patients With Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Darolutamide in Addition to Standard Androgen Deprivation Therapy and Docetaxel in Metastatic Hormone-Sensitive Prostate Cancer
Acronym: ARASENS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17777; 2015-002590-38 (EudraCT Number)
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Results first posted 2023-02-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: interventions — darolutamide; Androgen Antagonists; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAY1841788 /darolutamide (ODM-201)+standard ADT+Docetaxel (Experimental): Co-administration of BAY 1841788 / darolutamide (ODM-201), standard ADT and docetaxel
  Interventions: Drug: BAY1841788 / darolutamide (ODM-201); Drug: Standard ADT (androgen deprivation therapy); Drug: Docetaxel
- Placebo + standard ADT + Docetaxel (Placebo Comparator): Co-administration of Placebo matching BAY 1841788 / darolutamide (ODM-201) tablets, standard ADT and docetaxel
  Interventions: Drug: Standard ADT (androgen deprivation therapy); Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: BAY1841788 / darolutamide (ODM-201) — 600mg (2 tablets of 300 mg) of darolutamide (ODM-201)/placebo twice daily with food, equivalent to a total a daily dose of 1200 mg in addition to standard ADT (luteinizing hormone releasing hormone (LHRH) agonist/antagonist or orchiectomy) and 6 cycles of docetaxel
  Arms: BAY1841788 /darolutamide (ODM-201)+standard ADT+Docetaxel
Drug: Standard ADT (androgen deprivation therapy) — As prescribed by the treating physician.
Drug: Docetaxel — As prescribed by the treating physician.
Drug: Placebo — Placebo matching darolutamide (ODM-201) tablets in appearance, bid orally with food, in addition to standard ADT (luteinizing hormone releasing hormone [LHRH] agonist/antagonist or orchiectomy) and 6 cycles of docetaxel.
  Arms: Placebo + standard ADT + Docetaxel

SUMMARY:
The purpose of the study is to assess the efficacy and safety of BAY1841788 (darolutamide (ODM-201)) in combination with standard androgen deprivation therapy (ADT) and docetaxel in patients with metastatic hormone sensitive prostate cancer.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter phase III study. The study population will consist of approximately 1300 subjects with metastatic hormone sensitive prostate cancer (mHSPC), who will be randomized (1:1 ratio) to receive 600 mg (2 x 300 mg tablets) of darolutamide (ODM-201)/placebo twice daily with food, equivalent to a total daily dose of 1200 mg, in addition to standard androgen deprivation therapy (ADT) and docetaxel. Subjects will be stratified at randomization for the extent of disease and for Alkaline Phosphatase levels. All subjects will be treated with ADT as standard therapy. Six cycles of docetaxel will be administered after randomization.

The subjects considered for inclusion in the study will have metastatic prostate cancer and will be candidates for ADT and docetaxel.

Treatment with darolutamide (ODM-201)/placebo will be administered until symptomatic progressive disease, change of antineoplastic therapy, unacceptable toxicity, until subject withdraws consent, withdrawal from the study at the discretion of the investigator or his/her designated associate(s), death, non-compliance, or if sponsor terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate.
* Metastatic disease
* Candidates for ADT and docetaxel.
* Started ADT with or without first generation anti androgen, but no longer than 12 weeks before randomization
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior treatment with: LHRH agonist/antagonists; second generation androgen receptor (AR) inhibitors such as enzalutamide, ARN-509, darolutamide (ODM-201), other investigational AR inhibitors; CYP17 enzyme inhibitor such as abiraterone acetate or oral ketoconazole as antineoplastic treatment for prostate cancer; chemotherapy or immunotherapy for prostate cancer prior to randomization.
* Treatment with radiotherapy/radiopharmaceuticals within 2 weeks before randomization.
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV)
* Had a prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e., pTis, pTa, and pT1) is allowed, as well as any other cancer for which treatment has been completed 5 years before randomization and from which the subject has been disease-free
* Gastrointestinal disorder or procedure which is expected to interfere significantly with absorption of study treatment.
* Inability to swallow oral medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (271):
- United States (55):
  - Chandler, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Duarte, California
  - Los Angeles, California
  - Palo Alto, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Gainesville, Florida
  - Miami Beach, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Billings, Montana
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Camden, New Jersey
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - The Bronx, New York
  - Concord, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Gahanna, Ohio
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Bala-Cynwyd, Pennsylvania
  - Camp Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - North Charleston, South Carolina
  - Dallas, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Milwaukee, Wisconsin
- Australia (4):
  - Sydney, New South Wales
  - Adelaide, South Australia
  - Kurralta Park, South Australia
  - Fitzroy, Victoria
- Belgium (7):
  - Wilrijk, Antwerpen
  - Antwerp
  - Brussels
  - Bruxelles - Brussel
  - Ghent
  - Gilly
  - Namur
- Brazil (10):
  - Cachoeiro de Itapemirim, Espírito Santo
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Natal, Rio Grande do Norte
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Rio de Janeiro
  - São Paulo
- Bulgaria (6):
  - Gabrovo
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Vratsa
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- China (22):
  - Hefei City, Anhui Province, Anhui
  - Beijing, Beijing Municipality
  - Xiamen, Fujian
  - Guangzhou, Guangdong
  - Shijiazhuang, Hebei
  - Zhengzhou, Henan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shengyang, Liaoning
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Yantai, Shandong
  - Xi’an, Shanxi
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Finland (7):
  - Helsinki, Uusimaa
  - Jyväskylä
  - Kuopio
  - Mikkeli
  - Oulu
  - Tampere
  - Turku
- France (20):
  - Angers
  - Besançon
  - Bordeaux
  - Brest
  - Cergy-Pontoise
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - Marseille
  - Montpellier
  - Nancy
  - Paris
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Saint-Grégoire
  - Saint-Herblain
  - Saint-Mandé
  - Strasbourg
  - Villejuif
- Germany (13):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Nürtingen, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Braunschweig, Lower Saxony
  - Rostock, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Jena, Thuringia
  - Berlin
- Israel (8):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Petah Tikva
  - Safed
  - Tel Aviv
  - Ẕerifin
- Italy (10):
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Trento, Trentino-Alto Adige
  - Cortona, Tuscany
  - Padua, Veneto
  - Verona, Veneto
- Japan (41):
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Asahi, Chiba
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Matsuyama, Ehime
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kita-gun, Kagawa-ken
  - Yokohama, Kanagawa
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Kashihara, Nara
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Sakai, Osaka
  - Suita, Osaka
  - Hamamatsu, Shizuoka
  - Shimotsuke, Tochigi
  - Utsunomiya, Tochigi
  - Bunkyo-Ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Koto-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka, Tokyo
  - Nakano-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Yonago, Tottori
  - Ube, Yamaguchi
  - Chiba
  - Fukuoka
  - Gifu
  - Kumamoto
  - Miyazaki
  - Nagasaki
  - Osaka
  - Tokushima
  - Wakayama
- Mexico (7):
  - Mexico City, Mexico City
  - México, D. F., Mexico City
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Querétaro City, Querétaro
  - Mazatlán, Sinaloa
  - Durango
- Netherlands (8):
  - Amsterdam
  - Dordrecht
  - Geleen
  - Hilversum
  - Hoofddorp
  - Nijmegen
  - The Hague
  - Tilburg
- Poland (8):
  - Lodz
  - Lublin
  - Poznan
  - Rybnik
  - Siedlce
  - Waliszew
  - Warsaw
  - Wroclaw
- Russia (6):
  - Barnaul
  - Chelyabinsk
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
- South Korea (7):
  - Gwangju, Gwangju Gwang''yeogsi
  - Guri-si, Gyeonggi-do
  - Seongnam-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daegu
  - Seoul
- Spain (9):
  - Sabadell, Barcelona
  - Palma de Mallorca, Illes Baleares
  - Málaga, Málaga
  - Barcelona
  - Cáceres
  - Córdoba
  - Lugo
  - Madrid
  - Valencia
- Sweden (5):
  - Gothenburg
  - Lund
  - Stockholm
  - Umeå
  - Uppsala
- Taiwan (5):
  - Kaohsiung City, Kaohsiung
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- United Kingdom (6):
  - Colchester, Essex
  - Romford, Essex
  - Middlesbrough, Yorkshire
  - Belfast
  - Glasgow
  - London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Hussain M, Tombal B, Saad F, Fizazi K, Sternberg CN, Crawford ED, Shore N, Kopyltsov E, Kalebasty AR, Bogemann M, Ye D, Cruz F, Suzuki H, Kapur S, Srinivasan S, Verholen F, Kuss I, Joensuu H, Smith MR. Darolutamide Plus Androgen-Deprivation Therapy and Docetaxel in Metastatic Hormone-Sensitive Prostate Cancer by Disease Volume and Risk Subgroups in the Phase III ARASENS Trial. J Clin Oncol. 2023 Jul 10;41(20):3595-3607. doi: 10.1200/JCO.23.00041. Epub 2023 Feb 16. PMID 36795843
- [Derived] Smith MR, Hussain M, Saad F, Fizazi K, Sternberg CN, Crawford D, Manarite J, Muslin D, Farrington T, Tombal B. Darolutamide and survival in metastatic, hormone-sensitive prostate cancer: a patient and caregiver perspective and plain language summary of the ARASENS trial. Future Oncol. 2022 Jul;18(21):2585-2597. doi: 10.2217/fon-2022-0433. Epub 2022 Jun 3. PMID 35656777
- [Derived] Smith MR, Hussain M, Saad F, Fizazi K, Sternberg CN, Crawford ED, Kopyltsov E, Park CH, Alekseev B, Montesa-Pino A, Ye D, Parnis F, Cruz F, Tammela TLJ, Suzuki H, Utriainen T, Fu C, Uemura M, Mendez-Vidal MJ, Maughan BL, Joensuu H, Thiele S, Li R, Kuss I, Tombal B; ARASENS Trial Investigators. Darolutamide and Survival in Metastatic, Hormone-Sensitive Prostate Cancer. N Engl J Med. 2022 Mar 24;386(12):1132-1142. doi: 10.1056/NEJMoa2119115. Epub 2022 Feb 17. PMID 35179323
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multinational study was conducted between 30-Nov-2016 First Participant First Visit and 11-Apr-2023 Last Participant Last Visit, in 23 countries/regions:
  Australia, Belgium, Brazil, Bulgaria, Canada, China, Czech Republic, Finland, France, Germany, Israel, Italy, Japan, Mexico, Netherlands, Poland, Russian Federation, South Korea, Spain, Sweden, Taiwan, UK, US
Pre-assignment Details: 1306 were randomly assigned in a 1:1 ratio to study treatment and 1305 were considered valid for efficacy analyses. A total of 1302 participants started treatment and were included to safety analyses.
Groups:
- Darolutamide (BAY1841788) + Docetaxel: Participants received darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg in addition to their standard treatment with docetaxel and androgen deprivation therapy (ADT).
  Docetaxel was administered for six cycles after randomization. The first cycle of docetaxel was administered within 6 weeks after start of study drug.
  ADT administration started ≤12 weeks before randomization.
- Placebo + Docetaxel: Participants received matching placebo to darolutamide in addition to their standard treatment with docetaxel and androgen deprivation therapy (ADT). Docetaxel was administered for six cycles after randomization. The first cycle of docetaxel was administered within 6 weeks after start of study drug.
  ADT administration started ≤12 weeks before randomization.
Period: Overall Study
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Started (Randomized: 1306 patients were randomized. One patient was excluded from analysis due to a GCP violation) | 651 | 654
Started Treatment | 651 | 651
Completed (Ongoing with treatment) | 0 | 0
Not Completed | 651 | 654
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 5 | 6
Not completed — Lost to Follow-up | 4 | 2
Not completed — Additional primary malignancy | 11 | 6
Not completed — Non-compliance with study drug | 14 | 12
Not completed — Adverse event associated with clinical disease progression | 24 | 26
Not completed — Withdrawal by Subject | 26 | 40
Not completed — Progressive disease - clinical progression | 131 | 276
Not completed — Progressive disease - radiological progression | 90 | 133
Not completed — Adverse event not associated with clinical disease progression | 49 | 27
Not completed — Death | 9 | 5
Not completed — Other | 287 | 118
Not completed — Study drug never administered | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 651 | 654 | 1305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 243 | 234 | 477
  >=65 years | 408 | 420 | 828
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 651 | 654 | 1305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 49 | 89
  Not Hispanic or Latino | 561 | 557 | 1118
  Unknown or Not Reported | 50 | 48 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants] — More than one race includes: "American Indian or Alaska Native", "Native Hawaiian or other Pacific Islander", and "Multiple"
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 231 | 245 | 476
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 26 | 28 | 54
    White | 345 | 333 | 678
    More than one race | 6 | 2 | 8
    Unknown or Not Reported | 43 | 46 | 89

OUTCOME MEASURES:

1. Primary Outcome: OS From Date of Randomization Until Death From Any Cause - Number of Events
Description: Overall survival (OS) was defined as the time from the date of randomization until death from any cause.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  Long-term (Survival) follow-up period: After Active follow-up, patients continued to be contacted approximately every 12 weeks by phone. The end of the Survival follow-up period was defined as when the patient died, was lost to follow-up, withdrew consent, or at the end-of-study.
Time Frame: From randomization of the first participant until death from any cause up to 25 OCT 2021 cut-off date 533 OS events were reached (approximate 59 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number of patients with event | 229 | 304
  Number of patients censored | 422 | 350
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — Hazard ratio < 1 indicates superiority of Darolutamide+docetaxel arm over Placebo+docetaxel arm. Hazard ratio and 95% CI was based on Cox Regression Model, stratified by EOD (Non-regional lymph nodes metastases only vs. Bone metastases with or without lymph node metastases vs. Visceral metastases with or without lymph node metastases or with or without bone metastases) and ALP (<ULN vs. >=ULN); p < 0.0001, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.675, 95% CI 2-sided [0.568 to 0.801]; One-sided p-value from log-rank test, stratified by EOD (Non-regional lymph nodes metastases only vs. Bone metastases with or without lymph node metastases vs. Visceral metastases with or without lymph node metastases or with or without bone metastases) and ALP (<ULN vs. >=ULN)

2. Secondary Outcome: Number of Participants With TEAEs
Description: TEAEs = Treatment-emergent adverse events, were defined as any event(s) arising or worsening after the first dose of darolutamide or placebo, until 30 days after the last dose of darolutamide or placebo administration.
Time Frame: From the first dose of darolutamide or placebo until 30 days after the last dose of darolutamide or placebo administration up to cut-off date for the final completion analysis 11 APR 2023 (approximately 77 months)
Population: The number of patients who started treatment is presented based on the randomized treatment assignment. One patient was randomized to the placebo+docetaxel arm but received at least one dose of darolutamide. This patient was included in the darolutamide+docetaxel arm in the analysis of all safety variables.
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 652 | 650
Participants
  Any TEAE | 649 | 643
  TESAE | 306 | 276
  TEAE leading to study drug dose modification | 172 | 112
  TEAE leading to permanent discontinuation of study drug | 90 | 69
  TEAE leading to docetaxel dose modification | 216 | 214
  TEAE leading to permanent discontinuation of docetaxel | 52 | 67
  Related to protocol-required procedure | 69 | 64
  Any study drug-related TEAE | 344 | 309
  Study drug-related TESAE | 30 | 24
  Study drug-related TEAE leading to study drug dose modification | 75 | 41
  Study drug-related TEAE leading to permanent discontinuation of study drug | 25 | 13

3. Secondary Outcome: Time to Castration-Resistant Prostate Cancer (CRPC) - Number of Events
Description: Time to castration-resistant prostate cancer was defined as the time from randomization to the first occurrence of one of the following events: PSA progression, Radiological progression by bone lesions, or Radiological progression by soft tissue and visceral lesions.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first occurrence of an CRPC event up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number of patients with event | 225 | 391
  Number of patients censored | 426 | 263

4. Secondary Outcome: Time to Castration-Resistant Prostate Cancer (CRPC) - Month
Description: Time to castration-resistant prostate cancer was defined as the time from randomization to the first occurrence of one of the following events: PSA progression, Radiological progression by bone lesions, or Radiological progression by soft tissue and visceral lesions.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | NA [NA to NA] — NA = Value cannot be estimated due to censored data | 19.1 [16.5 to 21.8]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.357, 95% CI 2-sided [0.302 to 0.421]; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Pain Progression - Number of Events
Description: Time to pain progression was defined as the time from randomization to the first date a patient experienced pain progression.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first occurrence of a pain progression event up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number of patients with event | 222 | 248
  Number of patients censored | 429 | 406

6. Secondary Outcome: Time to Pain Progression - Month
Description: Time to pain progression was defined as the time from randomization to the first date a patient experienced pain progression.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | NA [30.5 to NA] — NA = Value cannot be estimated due to censored data | 27.5 [22.0 to 36.1]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0058, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.792, 95% CI 2-sided [0.660 to 0.950]; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Symptomatic Skeletal Event Free Survival (SSE-FS) - Number of Events
Description: Symptomatic skeletal event-free survival (SSE-FS) was defined as the time from randomization to the first occurrence of an SSE or death from any cause, whichever occurred first.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first occurrence of an SSE event or death from any cause, whichever occurred first up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number of patients with event | 257 | 329
  Number of patients censored | 394 | 325

8. Secondary Outcome: Symptomatic Skeletal Event Free Survival (SSE-FS) - Month
Description: Symptomatic skeletal event-free survival (SSE-FS) was defined as the time from randomization to the first occurrence of an SSE or death from any cause, whichever occurred first.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | 51.2 [47.2 to NA] — NA = Value cannot be estimated due to censored data | 39.7 [36.0 to 42.3]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.609, 95% CI 2-sided [0.516 to 0.718]; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE) - Number of Events
Description: Time to the first SSE was defined as the time from randomization to the first occurrence of an SSE. Identical to the definition used for SSE-FS. Death was not considered as an event in this endpoint.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first occurrence of an SSE event up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number (%) of patients with event | 95 | 108
  Number (%) of patients censored | 556 | 546

10. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE) - Month
Description: Time to the first SSE was defined as the time from randomization to the first occurrence of an SSE. Identical to the definition used for SSE-FS. Death was not considered as an event in this endpoint.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | NA [NA to NA] — NA = Value cannot be estimated due to censored data | NA [NA to NA] — NA = Value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0081, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.712, 95% CI 2-sided [0.539 to 0.940]; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: Time to Initiation of Subsequent Antineoplastic Therapy - Number of Events
Description: Time to initiation of subsequent systemic antineoplastic therapy was defined as the time from randomization to the initiation of first subsequent systemic antineoplastic therapy.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the initiation of first subsequent systemic antineoplastic therapy up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number (%) of patients with event | 219 | 395
  Number (%) of patients censored | 432 | 259

12. Secondary Outcome: Time to Initiation of Subsequent Antineoplastic Therapy - Month
Description: Time to initiation of subsequent systemic antineoplastic therapy was defined as the time from randomization to the initiation of first subsequent systemic antineoplastic therapy.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | NA [NA to NA] — NA = Value cannot be estimated due to censored data | 25.3 [23.1 to 28.8]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — One-sided p-value; Hazard Ratio, log = 0.388, 95% CI 2-sided [0.328 to 0.458]; [other analysis details as in outcome 1, analysis 1]

13. Secondary Outcome: Time to Worsening of Disease-Related Physical Symptoms - Number of Events
Description: Time to worsening of disease-related physical symptoms was defined as the time from randomization to the first date a patient experienced an increase in disease-related physical symptoms based on the NCCN-FACT-FPSI-17 questionnaire.
  Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first increase in disease-related physical symptoms based on the NCCN-FACT-FPSI-17 questionnaire up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number (%) of patients with event | 351 | 308
  Number (%) of patients censored | 300 | 346

14. Secondary Outcome: Time to Worsening of Disease-Related Physical Symptoms - Month
Description: as for outcome 13
Time Frame: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | 19.3 [13.8 to 24.8] | 19.4 [15.4 to 27.6]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7073, Log Rank — One-sided p-value; Hazard Ratio (HR) = 1.043, 95% CI 2-sided [0.894 to 1.217]; [other analysis details as in outcome 1, analysis 1]

15. Secondary Outcome: Time to Initiation of Opioid Use for ≥7 Consecutive Days - Number of Events
Description: Time to the initiation of opioid use for ≥7 consecutive days was defined as the time fromrandomization to the date of the first opioid use for ≥7 consecutive days. Data of opioid use related to cancer pain was included in the analysis, and opioid use for non-malignant causes was excluded.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
Time Frame: From randomization of the first participant to the first opioid use for ≥7 consecutive days up to 25 OCT 2021 cut-off date approximately 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Participants
  Number of patients with event | 92 | 117
  Number of patients censored | 559 | 537

16. Secondary Outcome: Time to Initiation of Opioid Use for ≥7 Consecutive Days - Month
Description: Time to the initiation of opioid use for ≥7 consecutive days was defined as the time fromrandomization to the date of the first opioid use for ≥7 consecutive days. Data of opioid use related to cancer pain was included in the analysis, and opioid use for non-malignant causes was excluded.
  Treatment period: until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Months | NA [NA to NA] — NA = Value cannot be estimated due to censored data | NA [NA to NA] — NA = Value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0037, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.688, 95% CI 2-sided [0.523 to 0.906]; [other analysis details as in outcome 1, analysis 1]

17. Primary Outcome: OS From Date of Randomization Until Death From Any Cause - Month
Description: Treatment period: treatment was provided for all patients, twice daily, until disease progression (symptomatic progressive disease, change of systemic antineoplastic therapy), unacceptable toxicity, consent withdrawal, withdrawal at the discretion of the investigator, death, or non-compliance.
  Active follow-up visits from the discontinuation of the darolutamide or placebo treatment period for up to 1 year or until the patient could no longer travel to the clinic, died, was lost to follow-up, or withdrew informed consent and actively objected to collection of further data.
  Long-term (Survival) follow-up period: After Active follow-up, patients continued to be contacted approximately every 12 weeks by phone. The end of the Survival follow-up period was defined as when the patient died, was lost to follow-up, withdrew consent, or at the end-of-study.
  Median, percentile and other 95% CIs were computed using Kaplan-Meier estimates.
  NA = Value cannot be estimated due to censored data
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 651 | 654
Month | NA [NA to NA] — NA = Value cannot be estimated due to censored data | 48.9 [44.4 to NA] — NA = Value cannot be estimated due to censored data

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last administration, including adverse event of all-cause mortality at any time during the study, up to cut-off date for the final completion analysis 11 APR 2023 (approximately 77 months)
Description: Treatment-emergent AEs (TEAEs) were defined as any event(s) arising or worsening after the first dose of darolutamide or placebo, until 30 days after the last dose of darolutamide or placebo administration.
  Events causally related to treatment were considered as events causally related to either darolutamide / Docetaxel or Placebo / Docetaxel
  A total of 1305 patients were randomized for efficacy analysis, however 1302 patients only started treatment and were included to safety analyses.
Groups:
- Darolutamide (BAY1841788) + Docetaxel: Participants received darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg in addition to their standard treatment with docetaxel and androgen deprivation therapy (ADT). Docetaxel was administered for six cycles after randomization. The first cycle of docetaxel was administered within 6 weeks after start of study drug. ADT administration started <=12 weeks before randomization.
- Placebo + Docetaxel: Participants received matching placebo to darolutamide in addition to their standard treatment with docetaxel and androgen deprivation therapy (ADT). Docetaxel was administered for six cycles after randomization. The first cycle of docetaxel was administered within 6 weeks after start of study drug. ADT administration started <=12 weeks before randomization.
Arm/Group | Darolutamide (BAY1841788) + Docetaxel | Placebo + Docetaxel
All-Cause Mortality (participants affected / at risk) | 231/652 | 305/650
Serious Adverse Events (participants affected / at risk) | 306/652 | 276/650
Other Adverse Events (participants affected / at risk) | 636/652 | 634/650
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide (BAY1841788) + Docetaxel (N=652) | Placebo + Docetaxel (N=650)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 40 (40) | 39 (44)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 12 (17) | 14 (17)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bone marrow oedema syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 5 (6) | 1 (2)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal strangulation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Death (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2)
Hernia (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 15 (15)
Sudden death (General disorders) | 2 (2) | 3 (3)
General physical health deterioration (General disorders) | 1 (1) | 4 (4)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (4) | 2 (4)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Fournier's gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 16 (17) | 21 (22)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyomyositis (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 6 (6)
Septic shock (Infections and infestations) | 3 (3) | 2 (2)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (7) | 7 (11)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 3 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 0 (0)
Spinal cord infection (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
West Nile viral infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 4 (4)
Biopsy lymph gland (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 18 (24) | 10 (10)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 4 (4)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen abnormal (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (5)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (2) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 5 (7) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 7 (7)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 5 (5)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 3 (3) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (2) | 3 (3)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 6 (6)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 5 (8) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 6 (6)
Ureterolithiasis (Renal and urinary disorders) | 4 (5) | 1 (1)
Malignant urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 1 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Orchidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Bilateral orchidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Radical prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Product contamination (Product Issues) | 0 (0) | 1 (1)
Device deposit issue (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide (BAY1841788) + Docetaxel (N=652) | Placebo + Docetaxel (N=650)
Anaemia (Blood and lymphatic system disorders) | 185 (276) | 164 (227)
Neutropenia (Blood and lymphatic system disorders) | 62 (108) | 67 (103)
Lacrimation increased (Eye disorders) | 38 (40) | 43 (47)
Abdominal pain (Gastrointestinal disorders) | 36 (40) | 37 (40)
Constipation (Gastrointestinal disorders) | 149 (202) | 132 (162)
Diarrhoea (Gastrointestinal disorders) | 168 (229) | 157 (225)
Nausea (Gastrointestinal disorders) | 117 (150) | 134 (174)
Stomatitis (Gastrointestinal disorders) | 67 (87) | 57 (69)
Vomiting (Gastrointestinal disorders) | 53 (63) | 58 (69)
Asthenia (General disorders) | 71 (89) | 65 (83)
Fatigue (General disorders) | 222 (291) | 215 (287)
Malaise (General disorders) | 58 (78) | 67 (97)
Oedema peripheral (General disorders) | 175 (206) | 169 (194)
Pain (General disorders) | 30 (36) | 42 (48)
Pyrexia (General disorders) | 84 (104) | 83 (110)
Nasopharyngitis (Infections and infestations) | 46 (69) | 46 (56)
Upper respiratory tract infection (Infections and infestations) | 57 (73) | 46 (52)
Urinary tract infection (Infections and infestations) | 57 (91) | 63 (92)
Fall (Injury, poisoning and procedural complications) | 45 (64) | 33 (37)
Alanine aminotransferase increased (Investigations) | 99 (132) | 81 (103)
Aspartate aminotransferase increased (Investigations) | 87 (120) | 66 (84)
Neutrophil count decreased (Investigations) | 165 (432) | 151 (415)
Weight decreased (Investigations) | 27 (32) | 37 (37)
Weight increased (Investigations) | 116 (147) | 105 (130)
White blood cell count decreased (Investigations) | 155 (395) | 142 (360)
Blood alkaline phosphatase increased (Investigations) | 45 (53) | 43 (53)
Hyperglycaemia (Metabolism and nutrition disorders) | 77 (100) | 61 (74)
Decreased appetite (Metabolism and nutrition disorders) | 121 (157) | 86 (96)
Arthralgia (Musculoskeletal and connective tissue disorders) | 186 (270) | 173 (249)
Back pain (Musculoskeletal and connective tissue disorders) | 128 (154) | 121 (147)
Bone pain (Musculoskeletal and connective tissue disorders) | 80 (91) | 82 (96)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 51 (59) | 48 (54)
Myalgia (Musculoskeletal and connective tissue disorders) | 74 (103) | 65 (84)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 104 (148) | 78 (95)
Dizziness (Nervous system disorders) | 60 (69) | 52 (64)
Dysgeusia (Nervous system disorders) | 71 (88) | 80 (84)
Headache (Nervous system disorders) | 59 (72) | 49 (58)
Hypoaesthesia (Nervous system disorders) | 38 (44) | 29 (40)
Neuropathy peripheral (Nervous system disorders) | 77 (91) | 68 (72)
Paraesthesia (Nervous system disorders) | 42 (45) | 55 (66)
Peripheral sensory neuropathy (Nervous system disorders) | 65 (74) | 68 (72)
Insomnia (Psychiatric disorders) | 77 (85) | 80 (93)
Haematuria (Renal and urinary disorders) | 59 (73) | 36 (43)
Pollakiuria (Renal and urinary disorders) | 31 (33) | 43 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 87 (103) | 73 (83)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 (73) | 71 (78)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (50) | 34 (38)
Alopecia (Skin and subcutaneous tissue disorders) | 267 (268) | 264 (265)
Dry skin (Skin and subcutaneous tissue disorders) | 48 (54) | 35 (37)
Nail discolouration (Skin and subcutaneous tissue disorders) | 50 (51) | 52 (52)
Pruritus (Skin and subcutaneous tissue disorders) | 46 (54) | 52 (62)
Rash (Skin and subcutaneous tissue disorders) | 53 (64) | 45 (58)
Hypertension (Vascular disorders) | 86 (112) | 61 (72)
Hot flush (Vascular disorders) | 128 (141) | 122 (136)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer may recommend any changes to the Publication as deemed necessary for scientific purposes. If the Publication could hinder the ability to obtain patent protection for any Invention, Bayer may request a delay of the Publication for a reasonable period to be able to file the patent application, but not to exceed 6 months from the date publication is received for review. Bayer may request further delay in case the patent application has been filed and the priority application is incomplete.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT02799602/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT02799602/SAP_003.pdf